CLINICAL TRIAL: NCT05344768
Title: Personalised Exercise Training in Adolescents With Type 2 Diabetes for the Early Prevention of Beta Cell Dysfunction: Development of a New Algorithm to Integrate Clinical, Epigenomic and Machine Learning Models
Brief Title: Personalised Exercise Training in Adolescents With Type 2 Diabetes for the Early Prevention of Beta Cell Dysfunction
Acronym: PT4DEEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yasemin Çırak (Other)
Collaborators: Istinye University (Other)
Responsible Party: Sponsor-Investigator, Yasemin Çırak, Associate Professor, Head of Physiotherapy and Rehabilitation Department, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISU003
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise; Resistance Training

STUDY DESIGN:
Intervention Model Description: The patients included in the study will be divided into six groups; the control group (20 adolescents), the moderate continuous aerobic exercise training group (20 adolescents), the high-intensity interval training group (20 adolescents), the resistance exercise training group (20 adolescents), combination of moderate continuous aerobic exercise training with resistance exercise training group (20) and combination of high-intensity interval training with resistance exercise training (20 adolescents).
Who Masked: Investigator
Masking Description: Group assignments will seal in sequentially numbered opaque envelopes by a investigator who will not involved in data collection. Investigators who will make evaluations and outcome measurements will not know the distribution of the groups throughout the study and will be blind.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- control group (No Intervention): Patients in the control group will be asked to maintain their usual exercise and eating habits throughout the study. No intervention will be applied.
- moderate continuous aerobic exercise training group (Experimental): After the warm-up period (5 minutes), 35 minutes of continuous exercise training will be applied at 60% (moderate intensity) of the maximum oxygen consumption (VO2max) value obtained from cardiopulmonary exercise test with a bicycle ergometer. After the exercise training, the patients will be taken to a 5 minute cool-down period.
  Interventions: Other: aerobic exercise
- high-intensity interval training group (Experimental): After the warm-up period (5 minutes), the patient will be asked to cycle for 1 minute at a workload of 90% (high intensity) of the VO2max obtained from cardiopulmonary exercise test with a bicycle ergometer, and the patient will be asked to cycle for 2 minutes at a workload of 25% of the VO2max value. This cycle will be repeated 10 times. The patient will then be placed in a 5 minute cool-down period.
  Interventions: Other: high-intensity interval exercise training
- resistance exercise training group (Experimental): It will be planned as 3 sets of 10 repetitions resistance exercises with 50% of 1 maximum repetition. Exercises will be performed on chest press, pectoral, pulley, hip abductor and adductor, leg press, cable biceps curl, triceps push down, shoulder press, abdominal crunch machines. The program will be created with a rest period of 3 minutes between sets, 10 minutes of stretching before the exercise and 10 minutes of stretching and cooling exercises after the exercise.
  Interventions: Other: resistance exercise training
- combination of moderate continuous aerobic exercise training with resistance exercise training group (Experimental): The combination of moderate continuous aerobic exercise training with resistance exercise training will be applied to the patients.
  Interventions: Other: aerobic exercise; Other: resistance exercise training
- combination of high-intensity interval training with resistance exercise training (Experimental): The combination of high-intensity interval training with resistance exercise training will be applied to the patients.
  Interventions: Other: high-intensity interval exercise training; Other: resistance exercise training

INTERVENTIONS:
Other: aerobic exercise — Moderate intensity aerobic exercise training will be applied.
  Arms: combination of moderate continuous aerobic exercise training with resistance exercise training group; moderate continuous aerobic exercise training group
Other: high-intensity interval exercise training — High-intensity interval exercise training will be applied.
  Arms: combination of high-intensity interval training with resistance exercise training; high-intensity interval training group
Other: resistance exercise training — resistance exercise training will be applied
  Arms: combination of high-intensity interval training with resistance exercise training; combination of moderate continuous aerobic exercise training with resistance exercise training group; resistance exercise training group

SUMMARY:
Exercise training is a key component in the prevention and treatment of various chronic diseases such as Type 2 diabetes (T2DM). Adaptations and effects that occur with exercise training differ according to exercise protocols. Most exercise interventions in T2DM base their results on HbA1c. Since the molecular and epigenetic effects of exercise training on β-cell function have not been fully revealed, the importance and effect of exercise training have not been fully understood.

The patients included in the study will be divided into six groups; the control group (20 adolescents), the moderate continuous aerobic exercise training group (20 adolescents), the high-intensity interval training group (20 adolescents), the resistance exercise training group (20 adolescents), combination of moderate continuous aerobic exercise training with resistance exercise training group (20) and combination of high-intensity interval training with resistance exercise training (20 adolescents). At the beginning of the study, demographic and physical characteristics of the patients will be recorded, and anthropometric and laboratory evaluations, pulmonary function test, measurement of respiratory muscle strength and endurance, measurement of peripheral muscle strength, evaluation of functional and aerobic capacity, measurement of physical activity levels and energy consumption, evaluation of the quality of life, epigenetic analysis, evaluation of β-cell function and biochemical structure of insulin will be done.

All patients will receive exercise training 3 days a week for 16 weeks. All measurements and evaluations will be made before starting exercise training and after 16 weeks of exercise training. As a result of the data obtained, it will be tried to objectively present which type of exercise intervention, at which doses and frequencies, will be more effective for patients with T2DM, with its effect on epigenetic factors.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a metabolic disease characterized by hyperglycemia due to insulin secretion or insufficiency in insulin function. In Type 2 diabetes (T2DM), the most common type of DM, high body mass index, unhealthy diet, reduced physical activity, an unfavorable intrauterine environment, and adverse genetic predisposition is among the risk factors. Over the past 20 years, the prevalence of T2DM among adolescents has increased several folds in the World.

Compared to adults with T2DM who develop secondary complications at a later age despite being insulin resistant for years, adolescents develop clinical T2DM and complications more rapidly and aggressively. Adolescents with T2DM have very poor treatment outcomes and a rapid decline in their glycemic control with the current treatment protocols. Early onset of T2DM and prolonged exposure to these metabolic abnormalities amplifies the long-term micro and macrovascular complications of these children. Also, according to the T2DM atlas of the International Diabetes Federation, T2DM will reach an epidemic level in the 2045 projection in adolescents and young people. Therefore, preventing the development of T2DM, slowing down the progression of the disease, stopping and treatment gaining great importance.

The core metabolic factors in the development of T2DM in adolescents include IR in the liver, muscle, adipose tissue, and eventual β-cell failure. However, the detailed molecular mechanisms related to the pathological process are not yet clear. Oxidative stress, which is expressed as disruption of oxidative balance, attacks healthy cells in the body and causes deterioration in their functions and structures. It has been reported that oxidative stress plays an important role both in the pathogenesis of T2DM and in the development of disease-related complications. Also another important factor for the development of T2DM is IR. IR is more pronounced by obesity and a sedentary lifestyle. Unlike their adult counterparts, children tend to overproduce insulin disproportionately in response to IR. Studies have shown that peripheral IR plays a significant role in the initiation of type 2 DM. Considering the role of oxidative stress and IR in the pathogenesis of T2DM and its effect on the development of disease-related complications, it is thought that exercise training may be beneficial in the prevention and/or treatment of T2DM. Therefore, it is very important to define the adaptation mechanisms that explain the oxidative stress preventive and therapeutic potential of exercise training.

Epigenetic processes have been associated with predisposition and progression to T2DM in response to various lifestyle factors or environmental exposures, including malnutrition, obesity, physical inactivity, stress, and toxins. Increasing evidence indicates that dynamic changes in the epigenome can occur within an individual's lifetime and that these changes can affect metabolic health. The molecular mechanisms governing the protective effects of exercise in T2DM are not yet fully understood. Several recent studies have shown that there are epigenetic modifications with exercise. Although there are in-vitro studies investigating the protective effects of different exercise protocols at the molecular level, no human studies are showing their epigenetic modifications.

Exercise training is a key component in the prevention and treatment of various chronic diseases such as T2DM. Adaptations and effects that occur with exercise training differ according to exercise protocols. Most exercise interventions in T2DM base their results on HbA1c. Since the molecular and epigenetic effects of exercise training on β-cell function have not been fully revealed, the importance and effect of exercise training have not been fully understood.

Considering the role of oxidative stress and inflammation, epigenetic changes in the pathogenesis of T2DM, and the development of disease-related complications, exercise training will be effective in the prevention and/or treatment of T2DM in young people. For this reason, with this project, the optimal exercise protocol will be determined to improve β-cell dysfunction, which will ensure the formation and protection of oxidative balance and reduce IR.

Personalised medicine aims to predict therapeutic response according to a personal profile that includes clinical, physiological and genetic data. So with this project, the development of epigenetic marker panels that will predict an individual's response to a particular exercise training protocol will contribute to revealing personalised epigenetic memory. Better knowledge of these connections will allow for the development of personalised exercise training regimens that will allow a person to achieve their training goals with maximum efficiency. Also this project aims to establish an artificial intelligence platform that brings together data from clinical research on the effects of different exercise training protocols with the purpose of identifying predictors. All results will be combined into a single data platform to develop predictive models for the treatment response. This data platform help to develop a decision support system for personalised exercise training in adolescents with T2DM.

The patients included in the study will be divided into six groups; the control group (20 adolescents), the moderate continuous aerobic exercise training group (20 adolescents), the high-intensity interval training group (20 adolescents), the resistance exercise training group (20 adolescents), combination of moderate continuous aerobic exercise training with resistance exercise training group (20) and combination of high-intensity interval training with resistance exercise training (20 adolescents). At the beginning of the study, demographic and physical characteristics of the patients will be recorded, and anthropometric and laboratory evaluations, pulmonary function test, measurement of respiratory muscle strength and endurance, measurement of peripheral muscle strength, evaluation of functional and aerobic capacity, measurement of physical activity levels and energy consumption, evaluation of the quality of life, epigenetic analysis, evaluation of β-cell function and biochemical structure of insulin will be done.

All patients will receive exercise training 3 days a week for 16 weeks. All measurements and evaluations will be made before starting exercise training and after 16 weeks of exercise training.

As a result of the data obtained, it will be tried to objectively present which type of exercise intervention, at which doses and frequencies, will be more effective for patients with T2DM, with its effect on epigenetic factors. In addition, determining an optimal non-pharmacological treatment method for a disease defined as an epidemic in the 2045 projection will contribute to the prevention of mortality and morbidity and the reduction of health expenditures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2DM,
* Being between the ages of 10-19,
* Body mass index (BMI) below 40 kg/m2,
* Being able to cooperate and walk for the exercise training and evaluation methods.

Exclusion Criteria:

* Having type 1 diabetes,
* Known lung disease,
* Have had any cardiac event or surgery in the last six months,
* Diabetes complications such as nephropathy, retinopathy and severe neuropathy,
* Being on insulin therapy,
* Having a known cancer disease,
* Having a known autoimmune, rheumatological disease,
* Having any known neuromuscular disease,
* Having other known endocrine disease other than T2DM,
* Existence of limitations and diseases that may affect exercise training.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Anthropometric Evaluation | 1-24 month
  The body composition of individuals will be evaluated using bioelectrical impedance analysis of five segmental regions: trunk, lower extremities, and upper extremities.
Body mass index | 1-24 month
  Body mass index (BMI) is a value derived from the mass (weight) and height of a person. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2, resulting from mass in kilograms and height in metres. The BMI score will be recorded.
Forced vital capacity | 1-24 month
  Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from lungs after taking the deepest breath possible. It's measured by spirometry , which is a common breathing test to check lung function.
Forced expiratory volume in the first second | 1-24 month
  The forced expiratory volume in 1 second (FEV1) is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration. Normally, at least 80% of the forced vital capacity (FVC) is exhaled in the first second.
The ratio of forced expiratory volume in the first second to the forced vital capacity | 1-24 month
  The ratio of forced expiratory volume in the first second to the forced vital capacity (FEV1/FVC) is a calculated ratio used in the diagnosis of obstructive and restrictive lung disease. It represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC). The result of this ratio is expressed as FEV1%. Normal values are approximately 75%.
Peak flow rate | 1-24 month
  The peak expiratory flow (PEF) is a person's maximum speed of expiration, as measured with a peak flow meter, a small, hand-held device used to monitor a person's ability to breathe out air.
Respiratory muscle strength and endurance test | 1-24 month
  In the evaluation of respiratory muscle strength, the patients' maximum inspiratory intraoral pressure (MIP) and maximum expiratory intraoral pressure (MEP) will be measured using a portable, electronic oral pressure measuring device, their values will be recorded in cmH2O.
Peripheral muscle strength test | 1-24 month
  As peripheral muscle strength, the strength of the shoulder abductor and adductor, shoulder flexor, extensor, elbow flexor and extensor muscles will be measured with a portable manual muscle strength measuring device.
Cardiopulmonary exercise test | 1-24 month
  Cardiopulmonary exercise test (KPET) will be performed with the measurement method (breath by breath) with each breath using the COSMED device.
Physical activity and energy consumption measurement | 1-24 month
  Physical activity levels will be evaluated with a three-dimensional accelerometer device (ActiGraph), which collects and stores movement information with microsensors.
Quality of life measurement | 1-24 month
  Quality of life will be assessed using the Diabetes-39 Quality of Life Scale (D-39). It is a disease-specific quality of life assessment scale developed to evaluate the quality of life of patients with diabetes.D-39 consists of 39 items and 5 domains (Diabetes control, Anxiety and worry, Social burden, Sexual functioning and Energy and mobility).Each item is scored between 1 and 7, the total score is 100, and high total scores indicate deteriorating quality of life.
Methylome analysis with next-generation sequencing | 1-24 month
  DNA sequences of bisulfite-converted samples will be sequenced by next generation sequencing, methylation and methylation patterns in CpG, CHG and CHH motifs on the promoter and other gene portions of the genes in the DNA obtained from each sample will be subjected to a genome-wide DNA methylation analysis using the relevant program. . Methylation scores will be calculated by comparing it with the genome before exercise. After performing the statistical analyzes, the methylation frequency in the CG, CHG and CHH sequences between the control and study groups will be directly related to the frequency and distribution of these sequences, in other words, whether there is a methylation effect will be tested statistically.
β-cell function analysis | 1-24 month
  C peptide level in the blood will be evaluated.C peptide level is based on blood sugar level. C peptide is a sign that your body is producing insulin. A low level indicates that the pancreas is producing little or no insulin.